CLINICAL TRIAL: NCT00498758
Title: The APOS System: Effects on Gait, Mobility and QOL in Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tasmc-07-ng-152-ctil
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-07

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Gait Disturbances; Mobility; Quality of life
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: APOS System - biomechanical wedge shoe

SUMMARY:
The purpose of this study is to evaluate the benefits of a biomechanical wedge system - The APOS system, for improving the stability of gait, mobility and quality of life in Parkinson's disease patients.

DETAILED DESCRIPTION:
Recently, a biomechanical wedge system was developed for gait and balance training among patients suffering from gait disorders. The APOS system (APOS Medical & Sports Technologies Ltd, Hertzeliya, Israel) applies special semispherical shoes, with individually adjusted implants, to improve age- and disease-related loss in muscle strength and neuromuscular control. The semispherical rubber devices that are placed on the soles of the shoes at the hind-foot and mid-foot can be moved medially, laterally, forwards and backwards. The system can be individually adjusted in order to optimally balance loading and re-train postural control during gait. An additional advantage of this treatment approach is the extraordinary compliance. The system is easily adjusted, maintained, and allows safe gait training.

After randomization, all subjects will be fitted with the APOS system, These shoes alter the dynamic balance during all gait cycle phases, adjusting the center of gravity and training postural control.

The precise location of the two wedges is adjusted individually by expert trainers using standardized protocols. Subjects in the intervention group will receive a proper wedge; subjects in the sham group will receive an almost flat wedge that lacks the proper biomechanical characteristics. However, both shoes and wedges will look similar. All subjects will be instructed to start gradually, with a goal of reaching 30 minutes of in-home walking while wearing the special training shoes. As an extra pre-caution, all subjects will be asked to walk with the shoes only in the presence of a caregiver, spouse or other family member during the first month. Before moving to more independent training, subjects will be checked for safety.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Stage 2-3 Hoehn & Yahr

Exclusion Criteria:

* Peripheral neuropathic pain
* Dementia
* Severe orthopaedic condition
* c.v.a
* Hearing or vision loss
* Usage of walking aid

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
gait characteristics | 3 monthes
Quality of life | 3 monthes
Mobility | 3 monthes

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, MD, Principal Investigator — Movement Disorders Unit - Tel Aviv Sourasky medical center